CLINICAL TRIAL: NCT02642731
Title: Kidney Biomarkers of Acute Kidney Injury in Patients With Knee Arthroplasty- a Pilot Study
Brief Title: Kidney Biomarkers of Acute Kidney Injury in Patients With Knee Arthroplasty
Acronym: dexpolvi
Status: Completed | Type: Observational
Sponsor: Kuopio University Hospital (Other)
Responsible Party: Principal Investigator, Merja Kokki, MD, PhD, Kuopio University Hospital
Other Study IDs: 2013-03-07
Record Dates: First submitted 2015-12-25; First posted 2015-12-30 (Estimated); Last update posted 2018-02-27 (Actual); Status verified 2018-02

CONDITIONS: Arthroplasty, Replacement, Knee; Acute Kidney Injury
Keywords: total knee arthroplasty; Kidney function; Renal markers
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma for measurement of renal markers Urine for measurement of renal markers
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients for elective TKA: patients with normal or near normal plasma creatinine who come for elective total knee arthroplasty

SUMMARY:
Sensitive renal markers have been studied abundantly in connection with open heart, liver and transplantation surgery; however in major orthopaedic surgery their use is anecdotal. The aim of the present study is to evaluate use of sensitive renal markers, NGAL (Neutrophil gelatinase associated lipocalin ), KIM-1 (Kidney injury molecule- 1), LFABP (liver-type fatty acid-binding protein), and IL-18 (interleukin -18), in patients coming for elective TKA (total knee arthroplasty) as a pilot study before large study concerning acute kidney injury in orthopaedic surgery.

DETAILED DESCRIPTION:
Acute renal deterioration is a serious adverse event in elective surgery. Serum creatinine based diagnostics of acute kidney injury may delay diagnosis and produce false negative results since serum creatinine is affected by diet, muscle mass, used hydration therapy. In recent times new markers have been developed and tested in order to find sensitive, fast and reliable marker of renal deterioration.

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* allergy to NSAIDs

Exclusion Criteria:

* no informed consent

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients coming to elective knee arthroplasty
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2013-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Renal function | time zero hours to 48 hours
  S-creatinine, Cystatin C, estimated GFR

SECONDARY OUTCOMES:
Concentraton of sensitive renal markers | time zero hours to 24 hours
  U-NGAL, P-NGAL, U-KIM-1, U-IL-18

CONTACTS AND LOCATIONS:
Overall Officials: Merja Kokki, MD, PhD, Principal Investigator — Kuopio University Hospital
Locations (1):
- Kuopio University Hospital, Kuopio, Northern Savonia, Finland

IPD SHARING:
Plan to Share IPD: No